CLINICAL TRIAL: NCT07093112
Title: Decoding Gut-Brain Biomarkers and Developing a Minimally Intrusive Gut Microbiome Sampling: Enhancing Cognitive Well-being in Athletes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Universidade do Extremo Sul Catarinense (UNESC) (Unknown); National Football League Players Association (NFLPA) (Unknown)
Responsible Party: Principal Investigator, Tatiana Barichello, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: HSC-MS-24-0876
Record Dates: First submitted 2025-05-27; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Athletic Performance; Gut Health

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Psychobiotic supplement (Experimental)
  Interventions: Dietary Supplement: Psychobiotic supplement
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Psychobiotic supplement — The psychobiotic supplement consists of Bifidobacterium lactis CCT 7858 and Lactobacillus rhamnosus CCT 7863, at a final concentration of 1 x 10^10 CFU/g (GABBIA® Biotechnology, Santa Catarina, Brazil).
  The intervention will be administered once daily for 90 days, spanning the pre-season and start-season phases with an interval and restarting for 90 days until the end-season phase.
  Arms: Psychobiotic supplement
Dietary Supplement: Placebo — The placebo consists of maltodextrin. The intervention will be administered once daily for 90 days, spanning the pre-season and start-season phases with an interval and restarting for 90 days until the end-season phase.
  Arms: Placebo

SUMMARY:
The objective of this study is to assess the impact of a psychobiotic supplement on the gut health, neurological markers, and behavior of younger soccer players over the soccer season.

ELIGIBILITY:
Inclusion Criteria:

* soccer player affiliated with Criciúma Esporte Clube (CEC)'s base in Criciúma, Santa Catarina, Brazil
* agree to participate voluntarily

Exclusion Criteria:

* athletes who withdraw from the study, cannot collect biological samples or answer the questionnaires during the pre-established times, and fail to take the capsules recommended in the study

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Recovery Process as Assessed by the Questionario de Estresse e Recuperacao para Atletas (RESTQ-Sport) - Stress Subscale | baseline, 30 days, 1 year
  The Questionário de Estresse e Recuperação para Atletas (RESTQ-Sport) assesses stress and recovery in athletes across 19 multidimensional scales: seven for general stress, five for general recovery, three for sports-specific stress, and four for sports-specific recovery. The RESTQ-Sport measures how well athletes recover from physical and mental stress over the previous three days and nights, providing a comprehensive understanding of their overall recovery status. The stress subscale score will be transformed into a percentage for a total score ranging from 0 to 100. A higher score on the stress subscale indicates a worse outcome (higher stress).
Recovery Process as Assessed by the Questionario de Estresse e Recuperacao para Atletas (RESTQ-Sport) - Recovery Subscale | baseline, 30 days, 1 year
  The Questionário de Estresse e Recuperação para Atletas (RESTQ-Sport) assesses stress and recovery in athletes across 19 multidimensional scales: seven for general stress, five for general recovery, three for sports-specific stress, and four for sports-specific recovery. The RESTQ-Sport measures how well athletes recover from physical and mental stress over the previous three days and nights, providing a comprehensive understanding of their overall recovery status. The recovery subscale score will be transformed into a percentage for a total score ranging from 0 to 100. A higher score on the recovery subscale indicates a better outcome (better recovery).
Preparation for Injury Prevention as Assessed by the Musculoskeletal Injury Readiness Questionnaire (MIR-Q) | baseline, 30 days, 1 year
  This questionnaire was developed for use with Brazilian athletes, particularly focusing on screening for musculoskeletal injury risks in various sports populations. One overall score will be reported, and the score will be transformed into a percentage for a total score ranging from 0 to 100. A higher score indicates a better outcome, suggesting that the athlete is more prepared for injury prevention.
Overtraining as assessed by the Overtraining Questionnaire | baseline, 30 days, 1 year
  The Overtraining Questionnaire measures overtraining syndrome in athletes, focusing on physical, psychological, social, and physiological factors, and it is designed to identify early signs of overtraining and prevent further progression of symptoms. The Brazilian adaptation will be used. The questionnaire is divided into six subscales: performance, psychological state, physiological responses, social factors, nutrition, and infection. One overall score will be reported, and the score will be transformed into a percentage for a total score ranging from 0 to 100. A higher score indicates a worse outcome, representing a higher risk or symptoms of overtraining.
Psychological distress as Assessed by the General Anxiety Disorder-7 (GAD-7) | baseline, 30 days, 1 year
  The Generalized Anxiety Disorder-7 (GAD-7) focusses on symptoms like excessive worry and difficulty controlling anxiety, as well as physical symptoms such as restlessness and fatigue. The GAD-7 was adapted for Brazilian Portuguese for use with the general adult population and has been validated for different age groups, including adolescents in Brazil. One overall score will be reported, and the score will be transformed into a percentage for a total score ranging from 0 to 100. A higher score indicates a worse outcome (greater anxiety).
Psychological distress as Assessed by the Patient Depression Questionnaire - Adolescents (PHQ-A) | baseline, 30 days, 1 year
  The Patient Health Questionnaire-9 (PHQ-9) measures the severity of depressive symptoms in clinical and non-clinical populations. It consists of nine items that assess the frequency of depressive symptoms over the past two weeks. The PHQ-9 was adapted for Brazilian Portuguese and validated among adults in the general population in Pelotas, Brazil. Each item is rated on a scale from 0 (not at all) to 3 (nearly every day), providing a total depression severity score. The score will be transformed into a percentage for a total score ranging from 0 to 100, and this will be reported. A higher score indicates a worse outcome (i.e., greater depressive symptoms).

SECONDARY OUTCOMES:
Psychological distress as Assessed by the Athletic Coping Skills Inventory - Brazilian Portuguese version (ACSI-25BR) | baseline, 30 days, 1 year
  The Athletic Coping Skills Inventory was developed to assess psychological coping skills in athletes. A Brazilian Portuguese version of the ACSI called the ACSI-25BR, which was adapted for Brazilian athletes, will be used. The ACSI is a multidimensional instrument, divided into seven subscales: coping with adversity, peaking under pressure, goal setting and mental preparation, concentration, freedom from worry, confidence and motivation, and coachability. The total score on these items reflects an athlete's overall coping resources. The total score will be transformed into a percentage for comparison (ranging from 0 to 100). A higher score indicates a better outcome, suggesting stronger coping skills.
Cognitive function as Indicated by Impulsivity as Assessed by the Delay Discounting Task (DD) | baseline, 30 days, 1 year
  The Delay Discounting (DD) Task measures impulsivity through repeated choices between a smaller, immediately available reward and a larger, delayed reward. A Brazilian Portuguese adaptation will be used. The k value will be reported. The k value is represents an individual's discount rate and is often used as a measure of behavioral impulsivity. The k value is obtained by the formula V=A/(1+kD) ), where V is the present value of the future reward, A is the reward amount, and D is the delay associated with the reward. The k value (discount rate) typically ranges from very low (around 0.00016) to high (around 0.25). A higher discount rate (k) (which indicates choosing smaller immediate rewards) indicates a worse outcome, suggesting higher impulsivity.
Cognitive function as Assessed by the Barkley Deficits in Executive Functioning Scale (BDEF) | baseline, 30 days, 1 year
  The Barkley Deficits in Executive Functioning Scale (BDEFS) assesses deficits in executive functioning in adults. It consists of 89 items that evaluate executive functioning across five domains: self-management of time, self-organization and problem-solving, self-restraint, self-motivation, and self-regulation of emotion. The BDEFS provides a comprehensive measure of the impact of executive function deficits on daily life, particularly in managing tasks, time, and emotions. The Brazilian Portuguese adaptation of the BDEFS will be used. The score will be transformed into a percentage for a total score ranging from 0 to 100. A higher score indicates a worse outcome, representing greater deficits in executive functioning.
Cognitive function as Assessed by the Trail Making Test (TMT) | baseline, 30 days, 1 year
  The Trail Making Test (TMT) assesses processing speed, cognitive flexibility, attention, and visual-motor speed. The time taken to complete the task will be reported and ranges from 0 to 5 minutes. A greater time indicates a worse outcome, reflecting slower cognitive processing speed.
Cognitive function as Assessed by the Verbal Fluency Test (VFT) | baseline, 30 days, 1 year
  The Verbal Fluency Test (VFT) assesses verbal memory, lexical retrieval, and cognitive flexibility, with a focus on both phonemic and semantic fluency. The test includes tasks that require participants to generate as many words as possible beginning with a specific letter (phonemic fluency) or generate as many words as possible from a given category (semantic fluency). The Brazilian Portuguese adaptation will be used. A total score will be reported, which is the number of correct words produced. A higher score indicates a better outcome, representing better verbal fluency and cognitive flexibility.
Cognitive function as Assessed by the Wechsler Adult Intelligence Scale®, Third Edition (WAIS-III) | baseline, 30 days, 1 year
  The Digits subtest from the Wechsler Adult Intelligence Scale, Third Edition (WAIS-III) consists of two parts: a forward task, where participants repeat a sequence of digits in the same order, and a backward task, where they repeat the sequence in reverse. The longest correctly repeated sequence is used to evaluate working memory capacity and cognitive load. The Brazilian Portuguese adaptation will be used. The score is based on the longest sequence of digits correctly recalled (0-14 forward and 0-12 backward). Total score will be reported and ranges from 0 to 28. A higher score indicates a better outcome, reflecting greater working memory capacity.
Childhood Trauma as Assessed by the Childhood Trauma Questionnaire (CTQ) | baseline, 30 days, 1 year
  The Childhood Trauma Questionnaire evaluates five types of childhood trauma: emotional abuse, physical abuse, sexual abuse, emotional neglect, and physical neglect. Each form of trauma is scored on a Likert scale, with higher scores indicating more severe trauma. The main outcomes help The questionnaire quantifies the impact of early life stress on later health and functioning. The Brazilian Portuguese adaptation will be used. The score will be transformed into a percentage for a total score ranging from 0 to 100. A higher score indicates a worse outcome, representing more severe childhood trauma.
Gastrointestinal Symptoms as Assessed by the Gastrointestinal Symptom Rating Scale (GSRS) | baseline, 30 days, 1 year
  The Gastrointestinal Symptom Rating Scale (GSRS) assesses the frequency and severity of gastrointestinal symptoms, particularly in patients with irritable bowel syndrome and peptic ulcer disease. The GSRS consists of 15 items that assess five domains: abdominal pain, reflux, indigestion, diarrhea, and constipation. The Brazilian Portuguese adaptation will be used. The score will be transformed into a percentage for a total score ranging from 0 to 100. A higher score indicates a worse outcome, reflecting more severe or frequent gastrointestinal symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Barichello, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Universidade do Extremo Sul Catarinense (UNESC), Criciúma, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: No